CLINICAL TRIAL: NCT01623297
Title: Cognitive Changes After Surgery in the Elderly: Does Minimally Invasive Surgery Influence the Incidence of Postoperative Cognitive Changes Compared to Open Colon Surgery?
Brief Title: Confusion in the Elderly After Colon Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: New York Hospital Queens (Other)
Collaborators: New York State Department of Health (Other Government)
Responsible Party: Principal Investigator, Mitchell Chorost, Principal Investigator, New York Hospital Queens
Other Study IDs: ECRIP
Record Dates: First submitted 2012-04-23; First posted 2012-06-19 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Confusion; Inflammation; Acute Phase Reaction; Surgery; Delirium
Keywords: Laparoscopy; Surgery; Acute Phase Reaction; Aged; Aged 80 and over; Confusion; Inflammation; Delirium
MeSH Terms: conditions — Confusion; Inflammation; Acute-Phase Reaction; Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples stored up to 7 months then expired and discarded
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Laparoscopic colon surgery: Patients over age 65 having laparoscopic colon resection for colonic adenocarcinoma
- Open colon surgery: Patients over age 65 having open colon resection for colonic adenocarcinoma

SUMMARY:
A study will be conducted to determine if there is any cognitive benefit in elderly patients having open versus minimally invasive colon cancer surgery.

DETAILED DESCRIPTION:
Cognitive changes in the elderly are common after surgery. It is not known if minimally invasive or laparoscopic surgery can prevent these changes. A study will be conducted on patients scheduled to have abdominal surgery. The patients will have cognitive evaluations before and after surgery. A small amount of blood, about 2 tablespoons, will be collected no more than 5 times in 6 months. The results will be analyzed to determine if there are changes between those having open surgery versus patients having laparoscopic or minimally invasive surgery, and if these changes coincide with cognitive changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients over age 65.0 years and in need of elective colon resection for adenocarcinoma

Exclusion Criteria:

* Inability to complete preoperative cognitive screening
* Inability to complete study in English since CANTAB is timed and not validated with interpreters
* Emergency surgery
* Depression or psychiatric comorbidity
* Pre-existing dementia
* Previous cerebrovascular accident or "stroke"
* Previous myocardial infarction
* Cardiac ejection fraction below 55%
* Propranolol, metoprolol or other betablocker use
* Digoxin, procainamide, or amiodarone use
* Calcium channel blocker use
* History of vascular surgery or arterial vascular disease
* History of alcohol dependence
* Lovastatin or other HMG-CoA reductase inhibitor use
* Ace inhibitor use
* Neuroendocrine or catecholamine associated tumors
* Hypertension
* Diabetes
* Benzodiazepine use
* Dimenhydrinate or other medications to treat motion sickness
* Metaclopramide use

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients newly diagnosed with colon adenocarcinoma will be contacted after being scheduled for surgery at New York Hospital Queens.
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Confusion | 6 Months
  Confusion assessed by questionaires and cognitive testing

SECONDARY OUTCOMES:
degree of inflammation | 6 Months
  5 separate blood draws
presence of electrolyte imbalance | 6 months
  5 separate blood draws
pituitary-thyroid axis disruption | 6 months
  5 separate blood draws
liver function tests | 6 months
  5 separate blood draws
nutritional status | 6 months
  5 separate blood draws

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell I Chorost, MD, Principal Investigator — New York Hospital Queens
Locations (1):
- New York Hospital Queens, Flushing, New York, United States

REFERENCES:
- [Background] Jemal A, Siegel R, Xu J, Ward E. Cancer statistics, 2010. CA Cancer J Clin. 2010 Sep-Oct;60(5):277-300. doi: 10.3322/caac.20073. Epub 2010 Jul 7. PMID 20610543
- [Background] Dyer CB, Ashton CM, Teasdale TA. Postoperative delirium. A review of 80 primary data-collection studies. Arch Intern Med. 1995 Mar 13;155(5):461-5. doi: 10.1001/archinte.155.5.461. PMID 7864702
- [Background] Juliebo V, Bjoro K, Krogseth M, Skovlund E, Ranhoff AH, Wyller TB. Risk factors for preoperative and postoperative delirium in elderly patients with hip fracture. J Am Geriatr Soc. 2009 Aug;57(8):1354-61. doi: 10.1111/j.1532-5415.2009.02377.x. Epub 2009 Jul 2. PMID 19573218
- [Background] Ansaloni L, Catena F, Chattat R, Fortuna D, Franceschi C, Mascitti P, Melotti RM. Risk factors and incidence of postoperative delirium in elderly patients after elective and emergency surgery. Br J Surg. 2010 Feb;97(2):273-80. doi: 10.1002/bjs.6843. PMID 20069607
- [Background] Rolfson DB, McElhaney JE, Rockwood K, Finnegan BA, Entwistle LM, Wong JF, Suarez-Almazor ME. Incidence and risk factors for delirium and other adverse outcomes in older adults after coronary artery bypass graft surgery. Can J Cardiol. 1999 Jul;15(7):771-6. PMID 10411615
- [Background] Roach GW, Kanchuger M, Mangano CM, Newman M, Nussmeier N, Wolman R, Aggarwal A, Marschall K, Graham SH, Ley C. Adverse cerebral outcomes after coronary bypass surgery. Multicenter Study of Perioperative Ischemia Research Group and the Ischemia Research and Education Foundation Investigators. N Engl J Med. 1996 Dec 19;335(25):1857-63. doi: 10.1056/NEJM199612193352501. PMID 8948560
- [Background] Layne OL Jr, Yudofsky SC. Postoperative psychosis in cardiotomy patients. The role of organic and psychiatric factors. N Engl J Med. 1971 Mar 11;284(10):518-20. doi: 10.1056/NEJM197103112841003. No abstract available. PMID 5100723
- [Background] Dimsdale JE, Newton RP, Joist T. Neuropsychological side effects of beta-blockers. Arch Intern Med. 1989 Mar;149(3):514-25. PMID 2563932
- [Background] Schubert DS, Gabinet L, Hershey LA. Psychosis induced by sustained-release procainamide. Can Med Assoc J. 1984 Nov 15;131(10):1188, 1190. No abstract available. PMID 6498664
- [Background] Trohman RG, Castellanos D, Castellanos A, Kessler KM. Amiodarone-induced delirium. Ann Intern Med. 1988 Jan;108(1):68-9. doi: 10.7326/0003-4819-108-1-68. No abstract available. PMID 3337520
- [Background] Binder EF, Cayabyab L, Ritchie DJ, Birge SJ. Diltiazem-induced psychosis and a possible diltiazem-lithium interaction. Arch Intern Med. 1991 Feb;151(2):373-4. PMID 1899553
- [Background] Bohner H, Hummel TC, Habel U, Miller C, Reinbott S, Yang Q, Gabriel A, Friedrichs R, Muller EE, Ohmann C, Sandmann W, Schneider F. Predicting delirium after vascular surgery: a model based on pre- and intraoperative data. Ann Surg. 2003 Jul;238(1):149-56. doi: 10.1097/01.sla.0000077920.38307.5f. PMID 12832977
- [Background] Dasgupta M, Dumbrell AC. Preoperative risk assessment for delirium after noncardiac surgery: a systematic review. J Am Geriatr Soc. 2006 Oct;54(10):1578-89. doi: 10.1111/j.1532-5415.2006.00893.x. PMID 17038078
- [Background] Marcantonio ER, Goldman L, Mangione CM, Ludwig LE, Muraca B, Haslauer CM, Donaldson MC, Whittemore AD, Sugarbaker DJ, Poss R, et al. A clinical prediction rule for delirium after elective noncardiac surgery. JAMA. 1994 Jan 12;271(2):134-9. PMID 8264068
- [Background] Redelmeier DA, Thiruchelvam D, Daneman N. Delirium after elective surgery among elderly patients taking statins. CMAJ. 2008 Sep 23;179(7):645-52. doi: 10.1503/cmaj.080443. PMID 18809895
- [Background] Vgontzas AN, Kales A, Bixler EO, Manfredi RL, Tyson KL. Effects of lovastatin and pravastatin on sleep efficiency and sleep stages. Clin Pharmacol Ther. 1991 Dec;50(6):730-7. doi: 10.1038/clpt.1991.213. PMID 1752118
- [Background] Lewis WH. Iatrogenic psychotic depressive reaction in hypertensive patients. Am J Psychiatry. 1971 Apr;127(10):1416-7. doi: 10.1176/ajp.127.10.1416. No abstract available. PMID 5549939
- [Background] Norkiene I, Ringaitiene D, Misiuriene I, Samalavicius R, Bubulis R, Baublys A, Uzdavinys G. Incidence and precipitating factors of delirium after coronary artery bypass grafting. Scand Cardiovasc J. 2007 Jun;41(3):180-5. doi: 10.1080/14017430701302490. PMID 17487768
- [Background] Dubois MJ, Bergeron N, Dumont M, Dial S, Skrobik Y. Delirium in an intensive care unit: a study of risk factors. Intensive Care Med. 2001 Aug;27(8):1297-304. doi: 10.1007/s001340101017. PMID 11511942
- [Background] Brown JH, Sigmundson HK. Delirium from misuse of dimenhydrinate. Can Med Assoc J. 1969 Dec 13;101(12):49-50. No abstract available. PMID 5362300
- [Background] Morgan DH. Neuro-psychiatric problems of cardiac surgery. J Psychosom Res. 1971 Mar;15(1):41-6. doi: 10.1016/0022-3999(71)90072-9. No abstract available. PMID 5576344
- [Background] Briggs W, Ruppert D. Assessing the skill of yes/no predictions. Biometrics. 2005 Sep;61(3):799-807. doi: 10.1111/j.1541-0420.2005.00347.x. PMID 16135031
- [Background] Briggs WM, Zaretzki R. The Skill Plot: a graphical technique for evaluating continuous diagnostic tests. Biometrics. 2008 Mar;64(1):250-6; discussion 256-61. doi: 10.1111/j.1541-0420.2007.00781_1.x. PMID 18304288
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204